CLINICAL TRIAL: NCT02307110
Title: A Cross Sectional Study Assessing the Prevalence of Different Stages of Diabetic Retinopathy and Diabetic Macular Edema Among Type 1 Diabetic Patients Treated With Long-term Intensified Insulin Therapy
Brief Title: Prevalence of DRP and DME Among Type 1 Diabetics Treated With Long-term Intensified Insulin Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vista Klinik (Other)
Collaborators: University Hospital, Basel, Switzerland (Other)
Responsible Party: Principal Investigator, Dr. med. Katja Hatz, Prof. Dr. Christian Pruente, Vista Klinik
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DRP-2010-02
Record Dates: First submitted 2014-11-25; First posted 2014-12-04 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2018-01

CONDITIONS: Insulin-Dependent Diabetes Mellitus 1
Keywords: Diabetes Mellitus 1; long-term intensified insulin therapy; diabetic retinopathy; diabetic macular edema
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetic Retinopathy | interventions — Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 arm study (Other): cross-sectional observation
  Interventions: Other: cross-sectional observation

INTERVENTIONS:
Other: cross-sectional observation — cross-sectional opthalmic examination
  Other Names: observational study.

SUMMARY:
This study is designed to evaluate the prevalence of different stages of diabetic retinopathy and diabetic macular edema among patients suffering from type 1 diabetes (DM 1) for 5 to 25 years and have been treated with intensified insulin therapy aiming near-normal blood glucose levels for the whole duration of disease.

Prevalence of different stages of diabetic retinopathy and diabetic macular edema is assessed using the modified Airlie House classification and the Early Treatment Diabetic Retinopathy Study (ETDRS) retinopathy severity scheme. Results of this study will provide the basis for designing further studies as well as staging and screening guidelines for diabetic retinopathy/diabetic macular edema.

DETAILED DESCRIPTION:
Purpose: This study is designed to evaluate the prevalence of different stages of diabetic retinopathy and diabetic macular edema among patients suffering from type 1 diabetes for 5 to 25 years and have been treated with intensified insulin therapy aiming near-normal blood glucose levels for the whole duration of disease.

Objectives: The primary objective is to examine the prevalence (percentages) of the stages of diabetic retinopathy (DR) and diabetic macular edema (DME) within one cross-sectional examination. Key secondary/exploratory objectives are the prevalence (percentages) of the stages of diabetic macular edema (DME), the means of individual average 5year-/10year-/15year-/20year-/25year-HbA1c value (%) as a measure for long-term glycemic control, the means of individual average 5year-/10year-/15year-/20year-/25year-blood pressure (mmHg) as a measure for long-term blood pressure control, mean BCVA score, mean contrast sensitivity score, mean NEI-VFQ 25 score (for further details see section Objectives).

Study design: Non-interventional cross-sectional investigator initiated study. The study will be conducted at Vista Klinik Binningen/Switzerland (ophthalmological evaluations) and the Department of Endocrinology of the University Hospital Basel/Switzerland (patient recruitment).

Study population: All patients with DM Type 1 with a least 5 years and maximum 25 years disease duration and intensified insulin therapy for the whole duration of disease, who are currently in follow-up for their DM1 at Department of Endocrinology of the University Hospital Basel/Switzerland. In order to prevent selection bias, patients will be screened for enrollment consecutively. For In-/exclusion criteria see section Eligibility.

Investigational and reference therapy: None.

Assessments:

* Visual acuity measurements using the ETDRS-like testing charts at a test distance of 4 meters
* Contrast sensitivity
* Ophthalmic examinations (slit lamp exam with fundus biomicroscopy, intraocular pressure)
* High resolution optical coherence tomography (Spectralis-OCT)
* Stereoscopic fundus photography
* Fluorescein angiography
* NEI-VFQ 25 (25-item National Eye Institute Vision Function Questionnaire)

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients >18 years of age who have signed an informed consent
* Patients with type 1 diabetes mellitus diagnosed between 5 and 25 years prior to screening who were on intensified insulin therapy (multiple daily insulin injections or insulin pump) from the beginning of the disease

Exclusion Criteria:

* Patients with hypertension and a change in antihypertensive treatment within 2 months pre-enrollment should not be enrolled unless blood pressure is maintained for at least 1 month below 160/100 mm Hg by antihypertensive treatment
* Patients with a history of chronic renal failure requiring dialysis or kidney transplantation if there is a risk for the patient to perform fluorescein angiography (discretion of the endocrinological investigator)
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (>5 mIU/ml)
* History of allergy to fluorescein
* Inability to obtain fundus photographs, fluorescein angiograms or OCT images of sufficient quality to be analyzed and graded
* Inability to comply with study procedures

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2010-08 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
prevalence (percentages) of the stages of diabetic retinopathy (DR) | one cross-sectional examination only

SECONDARY OUTCOMES:
prevalence (percentages) of the stages of diabetic macular edema (DME) | one cross-sectional examination only
  The outcome is evaluated for different patient groups relating to the duration of DM1 disease (5-10 years, 11-15 years, more than 15 years).
means of individual average 5year-/10year-/15year-/20year-/25year-HbA1c value (%) | 5year-/10year-/15year-/20year-/25year
  as a measure for long-term glycemic control
the means of individual average 5year-/10year-/15year-/20year-/25year-blood pressure (mmHg) | 5year-/10year-/15year-/20year-/25year
  as a measure for long-term blood pressure control
mean BCVA score | one cross-sectional examination only
  The outcome is evaluated for different patient groups relating to the duration of DM1 disease (5-10 years, 11-15 years, more than 15 years).
mean contrast sensitivity score | one cross-sectional examination only
  The outcome is evaluated for different patient groups relating to the duration of DM1 disease (5-10 years, 11-15 years, more than 15 years).
mean NEI-VFQ 25 score | one cross-sectional examination only
  The outcome is evaluated for different patient groups relating to the duration of DM1 disease (5-10 years, 11-15 years, more than 15 years).

CONTACTS AND LOCATIONS:
Overall Officials: Katja Hatz, MD, Principal Investigator — Vista Klinik Binningen
Locations (1):
- Vista Klinik, Binningen, Switzerland

REFERENCES:
- [Derived] Hatz K, Minder AE, Lehmann R, Drescher T, Gerendas B, Schmidt-Erfurth U, Kaider A, Pruente C, Zulewski H. The prevalence of retinopathy in patients with type 1 diabetes treated with education-based intensified insulin therapy and its association with parameters of glucose control. Diabetes Res Clin Pract. 2019 Feb;148:234-239. doi: 10.1016/j.diabres.2019.01.016. Epub 2019 Jan 23. PMID 30684505